CLINICAL TRIAL: NCT06654661
Title: Utilization of a 3D Printed Mechanical Balancer During Total Knee Arthroplasty (TKA)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-00350
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- TKA Patients (Experimental): TKA patients will undergo total knee replacement as part of standard of care. The 3D printed mechanical balancer will be used at one timepoint during surgery while the patient is under anesthesia during their scheduled TKA surgery.
  Interventions: Device: 3D-Printed Mechanical Balancer

INTERVENTIONS:
Device: 3D-Printed Mechanical Balancer — The 3D printed mechanical balancer is a surgeon-controlled handheld intraoperative tool used that provides a quantifiable measurement of force differences on the medial and lateral sides to guide achievement of a balanced knee. It will be used at one timepoint during scheduled TKA surgery while the patient is under anesthesia. Readings will be taken at 0, 45, and 90 degrees of flexion.

SUMMARY:
The aim of this study is to test a 3D-printed mechanical balancer in a clinical setting during surgery to further evaluate the utility of the device. This will be a pilot prospective study of 50 patients undergoing primary total knee arthroplasty. Surgeons will utilize the device intraoperatively in addition to the standard of care practices of mechanical balancing. It will not guide clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

* Surgical candidates undergoing primary TKA

Exclusion Criteria:

* Patient is unable to provide written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Measured Balance Value of the Medial Side of Knee during TKA | Day 1 (During TKA Procedure)
  Measured using the 3D-printed mechanical knee balancer.
Measured Balance Value of the Lateral Side of Knee during TKA | Day 1 (During TKA Procedure)
  Measured using the 3D-printed mechanical knee balancer.

SECONDARY OUTCOMES:
Range of Motion at Pre-Operative Visit | Baseline
Range of Motion at Post-Operative Visit | Up to Year 2 Post-Procedure
  Evaluated using chart review.
Cases of Revision Surgery | Up to Year 2
  Evaluated using chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Walker, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Daniel.waren@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Daniel.waren@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.